CLINICAL TRIAL: NCT03130751
Title: Mobile Self Management and Support for Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: BodiMojo, Inc. (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-002064
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application (Experimental)
  Interventions: Behavioral: Pocket Coach for AYA with Cancer

INTERVENTIONS:
Behavioral: Pocket Coach for AYA with Cancer — The Pocket Coach for AYA with Cancer is a psychosocial intervention to be delivered through a mobile platform. Intervention content is based on Mindfulness Based Stress Reduction (MBSR) and the Resilience in Illness Model [Dr. Joan E. Haase et al] and includes modules on relaxation, mindfulness, cognitions, and self-compassion.

SUMMARY:
This study is the user testing phase of a mobile application intervention which will be designed to promote positive coping skills, illness resilience, and social support, and to serve as a complement to patient-physician interactions in adolescents and young adults (AYA) with sarcoma. User testing will be conducted with a prototype of the app. Participants will be AYA ages 13-25 with sarcoma (N=16). Study participation involves the AYAs downloading and using the app for 30 days. During the 30 days, participants will interact with the app by inputting their current mood, receiving supportive feedback from the app, reading messages, and doing brief activities (such as relaxation activities, etc.). Participants will also participate in an online focus group focused around the user experience. Before and after the 30 days of user testing, participants will complete a few brief questionnaires about their behavior, how their symptoms affect their life, and how they receive support from others. These questions will take around 20 minutes to complete at each administration.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or self-reported (for participants 18+ years old) physician diagnosis of sarcoma
2. Daily use of a smartphone (iOS, Android, or Windows) or tablet
3. Current Facebook account that participant can use to participate in the focus group (or, be willing to create a Facebook account for this purpose).
4. Able and willing to give informed assent and comply with study requirements
5. For patients aged 13-17 years, have one caregiver willing and able to participate in the study
6. Able to read and speak English

Exclusion Criteria:

1. Patients that are not able to participate in the study due to their medical condition and/or treatment regimen, as determined by the patients' treating oncologist in conjunction with patients' family members
2. Inability to provide informed assent/permission/consent
3. Inability to read, speak, and understand English

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | 30 days (from day 1 through day 30 of the 30-day intervention period)
  Determined by the number of days participants use the program. Program usage will be assessed on the back end of the technology platform, which tracks how often each participant opens the app and uses any of the features. Intervention will be deemed feasible if participants use the program on at least two thirds of the 30 days in the study period (i.e., 20 out of the 30 days).

SECONDARY OUTCOMES:
Change in level of mindfulness | Pre-intervention to post-intervention (a span of 30 days)
  Assessed by the change in the total score on the Child and Adolescent Mindfulness Measure (CAMM) from pre-intervention to post-intervention. Calculated by subtracting the pre-intervention score from the post-intervention score. The CAMM is a 10-item measure whose total score can range from 0-40. Higher scores correspond to higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Pediatric Pain Program Research Offices, Los Angeles, California, United States

REFERENCES:
- [Derived] Donovan E, Martin SR, Seidman LC, Zeltzer LK, Cousineau TM, Payne LA, Knoll M, Weiman M, Federman NC. The Role of Social Media in Providing Support from Friends for Adolescent and Young Adult (AYA) Patients and Survivors of Sarcoma: Perspectives of AYA, Parents, and Providers. J Adolesc Young Adult Oncol. 2021 Dec;10(6):720-725. doi: 10.1089/jayao.2020.0200. Epub 2021 Apr 12. PMID 33844938
- [Derived] Donovan E, Martin SR, Seidman LC, Zeltzer LK, Cousineau TM, Payne LA, Trant M, Weiman M, Knoll M, Federman NC. A Mobile-Based Mindfulness and Social Support Program for Adolescents and Young Adults With Sarcoma: Development and Pilot Testing. JMIR Mhealth Uhealth. 2019 Mar 18;7(3):e10921. doi: 10.2196/10921. PMID 30882352